CLINICAL TRIAL: NCT03859115
Title: Effects of TENS on Myocardial Protection in Patients Undergoing AVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TENS_AVR
Record Dates: First submitted 2019-02-25; First posted 2019-03-01 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Myocardial Protection
Keywords: transcutaneous electrical nerve stimulation; sevoflurane; propofol; anesthesia; myocardial protection
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- preanesthesia-TENS (Active Comparator): Patients in preanesthesia-TENS group receive TENS for 30 minutes at one arm before anesthesia.
  Interventions: Procedure: TENS (transcutaneous electrical nerve stimulation)
- preanesthesia-sham (Sham Comparator): Patients in preanesthesia-sham group receive sham stimulation for 30 minutes at one arm before anesthesia.
  Interventions: Procedure: sham intervention
- sevoflurane-TENS (Experimental): Patients in sevoflurane-TENS group receive TENS for 30 minutes at one arm under sevoflurane anesthesia.
  Interventions: Procedure: TENS (transcutaneous electrical nerve stimulation)
- sevoflurane-sham (Active Comparator): Patients in sevoflurane-sham group receive sham stimulation for 30 minutes at one arm under sevoflurane anesthesia.
  Interventions: Procedure: sham intervention
- propofol-TENS (Experimental): Patients in propofol-TENS group receive TENS for 30 minutes at one arm under propofol anesthesia.
  Interventions: Procedure: TENS (transcutaneous electrical nerve stimulation)
- propofol-sham (Active Comparator): Patients in propofol-sham group receive sham stimulation for 30 minutes at one arm under propofol anesthesia.
  Interventions: Procedure: sham intervention

INTERVENTIONS:
Procedure: TENS (transcutaneous electrical nerve stimulation) — transcutaneous nerve stimulation with electrical pulse generation
  Arms: preanesthesia-TENS; propofol-TENS; sevoflurane-TENS
Procedure: sham intervention — sham stimulation without electrical pulse generation
  Arms: preanesthesia-sham; propofol-sham; sevoflurane-sham

SUMMARY:
Patients undergoing aortic valve replacement are randomized to receive TENS (transcutaneous electrical nerve stimulation) or sham stimulation at one arm for 30 min under various anesthetic conditions: no anesthesia (preanesthesia), sevoflurane or propofol anesthesia. Cardioprotective effects of TENS are compared through Langendorff rat heart perfusion system using plasma dialysate from patients.

DETAILED DESCRIPTION:
Patients undergoing aortic valve replacement are randomized to one of six groups: preanesthesia-TENS (transcutaneous electrical nerve stimulation), preanesthesia-sham, sevoflurane-TENS, sevoflurane-sham, propofol-TENS, propofol-sham. Patients receive TENS or sham stimulation (without electrical pulse generation) at one arm for 30 min under no anesthesia (preanesthesia) or sevoflurane or propofol anesthesia.

In all patients, blood samples are obtained before and after TENS or sham procedure to make plasma dialysate to perfuse rat hearts subjected to ischemia-reperfusion injury through Langendorff system.

Cardioprotective effects are determined by comparing infarct sizes of rat hearts perfused with human plasma dialysate, which reflects cardioprotective effects of TENS in human subjects. By comparing infarct size differences, the myocardial protective effects of TENS in various anesthetic conditions can be determined in human subjects undergoing aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing aortic valve replacement

Exclusion Criteria:

* co-medications: metformin, nitroglycerine, nicorandil
* discomfort at TENS or loss of intact skin
* uncontrolled hypertension or diabetes mellitus
* severely impaired renal or hepatic function
* peripheral vasculopathy or neuropathy
* did not consent to participate
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Infarct size after TENS | 30 minutes
  Infarct size of rat hearts perfused with dialysate after TENS compared with sham

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho YJ, Jung DE, Nam K, Bae J, Lee S, Jeon Y. Effects of transcutaneous electrical nerve stimulation on myocardial protection in patients undergoing aortic valve replacement: a randomized clinical trial. BMC Anesthesiol. 2022 Mar 9;22(1):68. doi: 10.1186/s12871-022-01611-x. PMID 35264104